CLINICAL TRIAL: NCT06768255
Title: A Multicenter, Randomized Controlled Trial of Abiraterone Acetate (II) Combined with ADT Versus Abiraterone Acetate Combined with ADT in Patients with Metastatic Castration-resistant Prostate Cancer
Brief Title: Phase III Study of Abiraterone Acetate (II) Versus Abiraterone Acetate in Patients with MCRPC
Acronym: mCRPC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ding-Wei Ye (Other)
Responsible Party: Sponsor-Investigator, Ding-Wei Ye, MD,PHD, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2411209-9; MA-PCa-III-011 (Other: Fudan University Shanghai Cancer Center)
Record Dates: First submitted 2024-12-30; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Abiraterone Acetate; MCRPC (metastatic Castration-resistant Prostate Cancer)
MeSH Terms: interventions — Abiraterone Acetate; BID protein, human; Androgen Antagonists; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Abiraterone acetate (II) +ADT+ prednisone (Experimental): Abiraterone acetate (II) (300 mg qd) + prednisolone (5mg bid) +ADT
  Interventions: Drug: Abiraterone Acetate (II)+ prednisolone (5mg bid) +ADT
- Abiraterone acetate +ADT+ prednisone (Active Comparator): Abiraterone acetate (1000 mg qd) + prednisolone (5mg bid) +ADT
  Interventions: Drug: Abiraterone acetate 1000 mg + prednisolone (5mg bid) +ADT

INTERVENTIONS:
Drug: Abiraterone Acetate (II)+ prednisolone (5mg bid) +ADT — Abiraterone Acetate（II）
  Arms: Abiraterone acetate (II) +ADT+ prednisone
Drug: Abiraterone acetate 1000 mg + prednisolone (5mg bid) +ADT — Abiraterone acetate 1000 mg
  Arms: Abiraterone acetate +ADT+ prednisone

SUMMARY:
Acetate abiraterone tablets (II) is a modified new drug launched in China, prepared using nanocrystal technology and supplemented with SNAC as an absorption enhancer, working together to promote the gastrointestinal absorption of Abiraterone, improve its oral bioavailability, and reduce its pharmacokinetic variability within individuals, as well as the impact of food on its pharmacokinetics. According to preliminary research results, the exposure to 300mg acetate abiraterone tablets (II) under fasting conditions is not less than the exposure to the original Zeke® 1000mg, and the food effect of acetate abiraterone tablets (II) is small, allowing for medication without dietary restrictions. The registration study uses steady-state serum testosterone levels as the primary pharmacodynamic indicator, comparing the efficacy of 300mg acetate Abiraterone tablets (II) and 1000mg Zeke® in mCRPC patients to be equivalent, with a safety advantage.This study is a non-inferior phase III, open-label, randomized controlled, multicenter trial. The study planned to enroll 400 mCRPC subjects and randomly assign them to the experimental group or the control group in a 1:1 ratio. The experimental group was treated with abiraterone acetate tablets (II.) combined with prednisone, and the control group was treated with abiraterone acetate tablets combined with prednisone, and the primary endpoints were PSA50 response rate and safety.To assess whether the efficacy (PSA50) of Abiraterone Acetate Tablets (II) is statistically non-inferior to that of Abiraterone Acetate Tablets, and whether there is a significant reduction in the incidence of grade 3 and above TEAEs.

ELIGIBILITY:
Inclusion Criteria:

1. Age≧ 18 years old, male;
2. Physical condition ECOG score 0~1 points;
3. Expected survival of at least 6 months;
4. Prostate adenocarcinoma confirmed by histological or cytological examination, and no diagnosis of neuroendocrine carcinoma or small cell carcinoma;
5. Ongoing luteinizing hormone-releasing hormone-releasing hormone (LHRHA) therapy (medical castration) or prior bilateral orchiectomy (surgical castration); Subjects who have not undergone bilateral orchiectomy must plan to maintain effective LHRHA therapy throughout the study;
6. Testosterone at castration level (≦50 ng/dL or 1.73 nmol/L) at screening;
7. Disease progression at the time of study enrollment. Disease progression is defined as the occurrence of one or more of the following 3 items while the subject is receiving castration therapy: (1) PSA progression, defined as PSA > 1 ng/mL with a PSA interval of 1 week, 2 consecutive episodes of >50% increase from the baseline value; In patients treated with flutamide or bicalutamide, PSA must also progress after discontinuation (≧ 4 weeks and ≧6 weeks, respectively); (2) disease progression as defined in RECIST 1.1; (3) Bone disease progression as defined by PCWG3 criteria, i.e., more than ≧2 new lesions found on bone scan;
8. Subjects who have been treated with one endocrine drug and/or one cytotoxic chemotherapeutic drug in the hormone-sensitive stage, such as novel androgen receptor antagonists (such as enzalutamide, apalutamide, ODM-201, revilutamide, HC-1119 and proxalutamide) or ADT (such as goserelin), etc., subjects who have been treated ≤with more than one treatment (bicalutamide for 4 weeks in the mCRPC stage can be included, and subjects who are on a triple regimen of new endocrine therapy combined with docetaxel can be included, Dual subjects with docetaxel in combination with ADT may be included);
9. Metastatic lesions confirmed by CT/MRI or radioactive bone scan (99mTc) imaging examination;
10. The functional level of the organ must meet the following requirements (no blood transfusion or hematopoietic growth factor therapy within 2 weeks prior to routine blood screening):

    * ANC≧1.5×10*9/L；
    * PLT≧100×10*9/L；
    * Hb≧80 g/L；
    * TBIL≦1.0×ULN；
    * ALT and AST ≦2.5×ULN;
    * BUN and Cr≦1.5×ULN.
11. As judged by the investigator, be able to comply with the test protocol;
12. Male subjects whose partner is a female of childbearing potential, should be surgically sterile or agree to use effective contraception during the trial and for at least 3 weeks after the last administration of abiraterone acetate tablets (Ecente) or abiraterone acetate (II), sperm donation is not allowed during the study;
13. Voluntarily participate in this clinical trial, understand the study procedures and have signed informed consent.

Exclusion Criteria:

1. Previous treatment with abiraterone acetate for prostate cancer;
2. Have received ≥2-line systemic drug therapy in the hormone-sensitive stage in the past;
3. Prior treatment with novel androgen receptor antagonists (such as enzalutamide, apalutamide, ODM-201, revilutamide, HC-1119 and proxalutamide), any cytotoxic chemotherapy drug therapy, molecularly targeted therapy (patients with HRR mutations who refuse or are unable to use PARP inhibitors can be enrolled) or immunotherapy in the mCRPC stage;
4. The washout period of any prior anti-tumor therapy (including radiotherapy, surgery, molecularly targeted therapy, immunotherapy, and first-generation androgen receptor antagonists) to the end of the randomization date of this study is < 4 weeks (except for the bicalutamide washout period < 6 weeks);
5. Participate in other drug clinical trials as subjects, and the last test drug administration is within 4 weeks from the randomization date of the drug in this study;
6. Plan to receive any other anti-tumor therapy during this trial;
7. Known untreated central nervous system (CNS) metastases. Patients with a history of surgery or radiotherapy for brain metastases, if the disease has been stable for at least 8 weeks after treatment prior to enrollment and corticosteroid-free for at least 2 weeks prior to enrollment;
8. Severe bone injury caused by tumor bone metastasis judged by the investigator, including severe bone pain with poor control, pathological fractures and spinal cord compression of important parts that occurred in the past 6 months or are expected to occur in the near future;
9. Presence of contraindications to prednisone (corticosteroid) use, such as active infection or other conditions;
10. Presence of any chronic condition requiring treatment with corticosteroids administered at doses greater than "prednisone 5 mg, BID";
11. Habitual constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease; Abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to the first dose of the drug; Those with abnormal gastrointestinal function, which may affect drug absorption as judged by the investigator;
12. Have a history of epilepsy, or have had diseases that can induce seizures within 12 months before C1D1 (including a history of transient ischemic attack, cerebral stroke, traumatic brain injury with impaired consciousness requiring hospitalization);
13. Uncontrolled hypertension. Subjects with a history of hypertension are allowed to participate in this study if they can effectively control their blood pressure through antihypertensive therapy;
14. Presence of active cardiac disease within 6 months prior to the randomization date of the study, including: severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, left ventricular ejection fraction <50%, and ventricular arrhythmias requiring medication;
15. Other malignant tumors within 5 years before the randomization date of the study (except for carcinoma in situ that has been in complete remission and malignant tumors that have been judged to have progressed slowly by the investigator);
16. Patients with active HBV or HCV infection (HBV virus copy number≧ 10*4 copies/mL, HCV virus copy number≧10*3 copies/mL);
17. History of immunodeficiency (including HIV test positive, other acquired and congenital immunodeficiency diseases) or organ transplantation;
18. Presence of inability to swallow, chronic diarrhea, intestinal obstruction or other factors affecting drug taking and absorption;
19. Known allergy or intolerance to abiraterone acetate or its excipients;
20. According to the judgment of the investigator, there are concomitant diseases (such as severe diabetes, peripheral neuropathy, thyroid diseases and psychiatric disorders, etc.) or any other conditions that seriously endanger the safety of the patient or affect the completion of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
PSA50 response rate | 24 months
  The main analysis of the PSA50 response rate will be performed based on the ITT set and the sensitivity analysis based on the PPS set. The number and percentage of participants achieving PSA50 response in each treatment group will be pooled, and the Clopper-Pearson method will be used to estimate the two-sided 95% confidence interval for PSA50 response rate in each treatment group. The difference in overall PSA50 response rate and rate stratification according to prior treatment modality (CAB vs. NHA vs. chemotherapy) between the two treatment groups will be pooled, and a two-sided 95% confidence interval for estimating the rate difference between groups using the Miettinen-Nurminen method will be used.

SECONDARY OUTCOMES:
ORR | 24 months
  RECIST1.1 criteria were used to assess tumor ORR, including cases of CR and PR. Definition of evaluable subjects: All subjects who meet the following criteria, i.e., presence of at least one measurable soft tissue lesion (according to criteria RECIST1.1) on baseline CT/MRI, at least 1 episode of study therapy, and at least 1 prior CT/MRI examination after initiation of study treatment. If the efficacy reaches CR and PR, the subject must be re-examined 4 weeks after the first evaluation. ORR is the number of subjects with an overall efficacy rating of CR or PR divided by the number of evaluable subjects.
PSA response rate | 24 months
  Evaluate the situation of PSA90 and PSA≤0.2ng/ml throughout the entire study period
The incidence of ALL Adverse events | 24 months
  Safety analysis will be based on the SS set, with the following data summarized descriptively separately based on the overall population and treatment group (only treatment-emergent adverse events [TEAEs] will be described): AEs, SAEs, ≥ Grade 3 AEs, Grade ≥3 SAEs, Drug-Related AEs, Drug-Related SAEs, AEs with an incidence of ≥5%, SAEs with an incidence of ≥5%, AEs leading to dose adjustments, AEs leading to discontinuation of treatment.
rPFS | 24 months
  rPFS (Radiographic Progression-Free Survival) time is defined as the time from the randomization date to the occurrence of radiographic disease progression (radiographic disease progression is based on the date of imaging examination, according to RECIST 1.1 and adjusted PCWG3 criteria) or death from any cause, calculated as the time of first occurrence.
OS | 24 months
  OS is defined as the time from the date of randomization to death from any cause.
Time to PSA progression | 24 months
  Time to PSA progression is defined as the time from randomization to first PSA progression;PSA progression is judged according to PCWG3 criteria, PSA level changes within the first 12 weeks of treatment are not included in this evaluation, and others are as follows:
  1. If PSA at the end of week 12 after randomization is lower than baseline, PSA progression is defined as an increase of ≥ 50% and an absolute increase of ≥ 1 ng/mL from the nadir level (nadir in PSA at the end of week 12 and thereafter);
  2. If PSA at the end of 12 weeks after randomization is not lower than baseline, PSA progression is defined as an increase from baseline ≥ 50% and an absolute increase ≥ 1 ng/mL;
  3. PSA progression on initial evaluation should be confirmed ≥ 3 weeks later.
Time to pain progression | 24 months
  Time to pain progression: the time from randomization to the date of 30% or greater improvement from baseline in pain severity score (using BPI-SF). or 2 consecutive assessments from the start of treatment to an interval ≥of 4 weeks to observe a 2-point increase from baseline in the most severe pain intensity of BPI-SF (scale point 3) or the time to initiation of chronic opioids, whichever occurs first.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Pudong New Area, China

IPD SHARING:
Plan to Share IPD: Undecided